CLINICAL TRIAL: NCT01145027
Title: Relations Among Cephalic Phase of Insulin Secretion, Body Composition, Dietary Intake and Microvascular Reactivity in Healthy Young Men
Brief Title: Cephalic Phase Insulin Secretion and Capillary Recruitment in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Caroline Buss, RD, MSc, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: do200812
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-06

CONDITIONS: Microvascular Function
Keywords: Capillary recruitment; Cephalic Phase of Insulin Secretion; Dietary Intake

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention)
- Sensorial Stimulus (Experimental): The sensorial stimulus will be a breakfast meal, with excellent presentation and aroma, composed by favorite food items previously related by the individual for this meal. The meal will not be offered for immediate intake, it will be placed in front of the volunteer for perception of the smell and taste, in order to trigger the cephalic phase of insulin secretion
  Interventions: Other: Breakfast tray

INTERVENTIONS:
Other: Breakfast tray — The sensorial stimulus will be a breakfast meal, with excellent presentation and aroma, composed by favorite food items previously related by the individual for this meal. The meal will not be offered for immediate intake, it will be placed in front of the volunteer for perception of the smell and taste.
  Arms: Sensorial Stimulus

SUMMARY:
Forty healthy volunteers will undergo two nailfold-videocapillaroscopy exams with a 10-minute interval between them, after an 10-h overnight fast in a temperature controlled room. The subjects will be randomized in two groups: one will receive a sensorial stimulus during the interval (stimulus group - SG) and the other will receive no stimulus (control group - CG). The sensorial stimulus will be a breakfast meal, with excellent presentation and aroma, composed by favorite food items previously related by the individual for this meal. The meal will not be offered for immediate intake, it will be placed in front of the volunteer for perception of the smell and taste.

Baseline microvascular parameters will be compared to the results after the interval. The investigators hypothesize that the SG will have greater capillary recruitment due to a possible effect of physiologically secreted insulin provoked by the sensorial stimulation (cephalic phase of insulin secretion).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Aged between 18 and 30 years
* BMI between 18.5 and 24.9 kg/m2

Exclusion Criteria:

* Diabetes mellitus, glucose intolerance or altered fasting glucose;
* Hypertension (Systolic pressure ≥ 130 mmHg and diastolic pressure ≥ 80 mmHg);
* HOMA-index ≥ 2.71
* Dyslipidemia
* Renal disease, coronary or peripheral vascular diseases, haematologic or hepatic diseases
* Smoking
* Chronic use of any medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
functional capillary density (number of perfused capillaries on the studied skin area) | up to 30 minutes

SECONDARY OUTCOMES:
cephalic phase of insulin secretion (the occurence of increase in markers of this phase, such as insulin, C-peptide and pancreatic polypeptide) | Up to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Buss, Master, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Laboratorio de Pesquisas Clinicas e Experimentais em Biologia Vascular, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Buss C, Kraemer-Aguiar LG, Maranhao PA, Marinho C, de Souza Md, Wiernsperger N, Bouskela E. Novel findings in the cephalic phase of digestion: a role for microcirculation? Physiol Behav. 2012 Feb 28;105(4):1082-7. doi: 10.1016/j.physbeh.2011.12.004. Epub 2011 Dec 14. PMID 22197630